CLINICAL TRIAL: NCT05073263
Title: Full Weightbearing Versus Partial Controlled Weightbearing During the First Six Weeks of Rehabilitation After Reconstruction of the Fibular Collateral Ligament: a Randomized Controlled Trial
Brief Title: Full Vs Partial Weightbearing During the First Six Weeks of Rehab. After Fibular Collateral Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Twin Cities Orthopedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RFL_FWB vs PWB-FCL
Record Dates: First submitted 2021-09-14; First posted 2021-10-11 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Knee Injuries
Keywords: fibular collateral ligament (FCL); anterior cruciate ligament (ACL)
MeSH Terms: conditions — Knee Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Partial weight -bearing for the first six weeks after surgery (Active Comparator): Partial weightbearing will be defined as 40% of the patient's body weight.
  Interventions: Other: Physical Therapy
- Full weight -bearing for the first six weeks after surgery (Experimental): If the patient is randomized to the full weightbearing group, the patient will be instructed about acceptable exercises and activities.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Patient is randomized to the weightbearing group the day after surgery.

SUMMARY:
This is a prospective randomized controlled trial with the purpose to determine if patients undergoing fibular collateral ligament (FCL) reconstruction alone or combined FCL and anterior cruciate ligament (ACL) reconstructions can safely begin full controlled weightbearing for the first six weeks after surgery.

DETAILED DESCRIPTION:
Patients will be randomly assigned to one of two rehabilitation protocols for the first six weeks post-surgery:

1. partial weightbearing
2. full controlled weightbearing

An immobilizer brace in extension will be used from post-operative day 0 through 13 and a CTi ligament knee brace (Össur Americas, Foothill Ranch, California) will be used from 14 to 42 days post-surgery to protect against side-to-side motion while weight bearing.

Specific Aims

1. Primary Aim: To determine if there is a difference in millimeters of varus gapping on anteroposterior (AP) stress radiographs at six months post-surgery between patients who are partial weight bearing versus full controlled weight bearing during the first six weeks of post-surgical rehabilitation. This distance will be compared to varus gapping measured on the contralateral uninjured control knee.
2. Secondary Aim: To determine if there is a difference in pain, edema, and range of motion, gait, quadriceps strength, and patient reported outcomes between groups.

The Investigators hypothesize that there will be no clinically significant difference (< 2 mm change) in varus gapping between the control and treatment groups. Results of this study will help to expedite return to pre-injury levels of activity and decrease adverse sequelae associated with non-weight bearing such as osteopenia, muscle atrophy, loss of ankle range of motion, and increased risk of deep vein thrombosis.

The current standard of care for FCL reconstruction is early controlled partial weight -bearing for the first six weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 14 years old, <60
* Reconstruction of FCL alone
* Combined FCL + ACL reconstructions
* Males or females
* Is willing and able to comply with the clinical trial plan and able to understand and sign the Patient Informed Consent Form.

Exclusion Criteria:

* < 14 years old, > 60
* Pregnant
* Revision FCL reconstructions
* Concurrent biceps femoris or lateral capsular repairs
* Concurrent PCL or MCL reconstructions
* Concomitant meniscus root or radial repair surgery with transtibial technique

Ages: 14 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Gapping (mm) measured on Standard of Care Varus stress radiographs | Pre-operative
  stress radiograph
Gapping (mm) measured Standard of Care Varus stress radiographs | 6 months post-surgery
  stress radiograph

SECONDARY OUTCOMES:
Numeric Pain Scale (NPS) (0-10 rating) | Baseline and 6 months
  Pain scale 0-100
Measurements by physical therapists (Edema, thigh circumference) | 4,7, and 10 months after surgery
  Measurements with tape
Measurements by physical therapists (Range of Motion) | 4,7, and 10 months after surgery
  Measurements with goniometer
Measurements by physical therapists (Quadriceps strength, gait analysis) | 4,7, and 10 months after surgery
  Measurements by biomechanics lab
Patient reported outcome scores | Baseline, 3 months, 6 months, 1 year
  Surveys: International Knee Documentation Committee (IKDC), Cincinnati Knee Rating System (Cincinnati), Knee injury and Osteoarthritis Outcome Score (KOOS), Tegner, Lysholm Knee Scoring Scale (Lysholm), and Veterans Rand 12 (VR-12) or Short Form-12 (SF-12) General Health Survey, lower extremity functional scale, Sports Medicine Questionnaire and survey/patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Robert F LaPrade, MD, PhD, Principal Investigator — Twin Cities Orthopedics
Locations (1):
- Twin Cities Orthopedics, Edina, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No